CLINICAL TRIAL: NCT04350996
Title: Application of a Wearable Alcohol Sensor for Prevention of Pancreatitis
Brief Title: Continuous Alcohol Monitoring for Pancreatitis
Acronym: CAMP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gillian Gresham, Assistant Professor, Cedars-Sinai Medical Center
Other Study IDs: STUDY00000526
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Pancreatitis; Alcohol Drinking
Keywords: Wearable technology; Remote monitoring; Pancreatitis; Continuous alcohol monitoring
MeSH Terms: conditions — Pancreatitis; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Continuous alcohol monitoring: Wearable BACtrack Skyn device
  Interventions: Other: Wearable alcohol sensor

INTERVENTIONS:
Other: Wearable alcohol sensor — BACtrack Skyn, is a novel transdermal blood alcohol sensor developed by BACtrack, a company established for police-grade breathalyzers, and winner of the Wearable Alcohol Biosensor Challenge sponsored National Institute on Alcohol Abuse and Alcoholism.

SUMMARY:
The purpose the research is to demonstrate the feasibility of using a transdermal alcohol sensing device (BACtrack Skyn), and to correlate biological and self-reported alcohol measures with the transdermal alcohol measures in patients with a history of pancreatitis. The results from this study will inform tailored, self-directed interventions for reducing alcohol consumption in persons with pancreatitis.

DETAILED DESCRIPTION:
Alcohol is the leading cause of recurrent acute and chronic pancreatitis, which greatly elevates the risk of pancreatic cancer. Reducing alcohol intake in patients with a history of alcoholic pancreatitis prevents progression of pancreatitis. Provider-based education on alcohol reduction has not translated to sustainable behaviors change, and more effective and scalable interventions are needed. Wearable alcohol sensors can empower patient-directed behavior change through real-time feedback on alcohol levels in the blood. BACtrack Skyn, the winner of NIAAA's Wearable Alcohol Biosensor Challenge, is a validated transdermal alcohol sensor that estimates blood alcohol concentration. In this pilot study, the investigators aim to (a) determine the feasibility and acceptability of using BACtrack Skyn to monitor changes in blood alcohol concentration among patients at risk for pancreatitis, (b) assess correlations between alcohol levels measured with BACtrack Skyn, breathalyzer, patient-reported alcohol consumption, and urine alcohol metabolite levels, (c) explore whether the use of a wearable alcohol sensor results in a decrease in alcohol consumption over a two-week period. Sixteen participants with known history of alcoholic pancreatitis will be assigned to wearing BACtrack Skyn for 2 weeks with the goal of not exceeding a blood alcohol concentration of 0.08%. Patient-reported drinking history, urine will be collected to correlate reported drinking levels and alcohol metabolic levels with the blood alcohol concentration readings in BACtrack Skyn. Findings from this study will be used as preliminary data to support and optimize subsequent grant applications and inform larger, randomized trials. The proposed study aligns closely with the mission of Cedars-Sinai and contributes to the growing body of research focusing on novel technologies for cancer prevention and control, as well as translational studies on alcoholic gastrointestinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years at the time of eligibility assessment
* History of at least one AP per Revised Atlanta Classification (20) within past 3 years from screening, which requires two of the following evidence of pancreatitis:
* Abdominal pain consistent with AP (acute onset of a persistent, severe, epigastric pain often radiating to the back)
* Serum lipase activity (or amylase activity) at least three times greater than the upper limit of normal
* Characteristic findings of AP on contrast-enhanced computed tomography (CECT), magnetic resonance imaging (MRI) or transabdominal ultrasonography
* Access to a mobile or portable device that has the capability to sync to the BACtrack sensor and internet connection for syncing purposes.

Exclusion Criteria:

* Pancreatitis presumed to be related to: gallstones, medication, trauma, autoimmune pancreatitis, post-ERCP pancreatitis, pancreatic ductal adenocarcinoma, suspected cystic neoplasm, neuroendocrine tumors, and other uncommon tumors.
* Episode of acute pancreatitis requiring hospitalization in the past 4 weeks.
* Current medical or psychiatric illnesses that in the investigator's opinion would compromise their ability to tolerate study procedures.
* Currently incarcerated.
* Known pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have acute or chronic pancreatitis without calcification and have alcohol consumption score of ≥ 3 as measured using the validated TWEAK scale.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled patients who wore the BACTrack sensor for at least 7 days within the 14-day period | up to 14 days
  Feasibility based on proportion of patients who wore the BACTrack sensor for at least 50% of study duration

SECONDARY OUTCOMES:
Acceptability of the BACtrack Skyn using the System Usability Scale (SUS) | 14 days
  SUS is a 10 item questionnaire, with 5 Likert-type response options (range 1(strongly disagree) to 5 (strongly agree)). Sensors will be deemed acceptable if ≥75% of the study population report an acceptability score of 68 or greater
Blood alcohol concentration (BACtrack breathalyzer) | up to 14 days
  Daily levels of estimated BAC using breathalyzer (continuous)
Patient-reported alcohol consumption | up to 14 days
  Number of alcoholic beverages each day
Urine alcohol consumption | 14 days
  Urine alcohol metabolite (ethyl glucuronide [EtG]) levels (continuous)
Patient-reported pain | up to 14 days
  Daily visual analog scale (range 0(low)-10 (high))

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No